CLINICAL TRIAL: NCT02773160
Title: Motor Learning for the Lumbar Spine Using Sensor-based Postural Feedback: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Annick Timmermans, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AcuteLearningEffects
Record Dates: First submitted 2016-01-11; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Non-specific Low Back Pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sensor-based postural feedback (Experimental): Subjects will receive visual feedback on a computer screen while practicing the motor control task. The feedback is based on information from from motion sensors that mointor the movements of the lumbar spine
  Interventions: Other: Sensor-based postural feedback
- Mirror Feedback (Experimental): Subjects will receive feedback from a mirror while practicing the motor control task
  Interventions: Other: Mirror feedback
- control group (Active Comparator): Subjects will receive no feedback while practicing the motor control task
  Interventions: Other: Control group

INTERVENTIONS:
Other: Sensor-based postural feedback — Motion tracking sensors will provide feedback to subjects during the learning phase of a motor control task
  Arms: Sensor-based postural feedback
Other: Mirror feedback — Subjects will receive feedback from a mirror during the learning phase of a motor control task
  Arms: Mirror Feedback
Other: Control group — Subjects will receive no feedback during the learning phase of a motor control task
  Arms: control group

SUMMARY:
A large subgroup of patients with chronic non-specific low back pain have motor control impairments. During motor control exercises, different forms of external feedback can be used to support training. This randomized controlled trial will investigate the effectiveness of different forms of external feedback during the learning phase of a motor control task for the lumbar spine in healthy subjects and patients with chronic non-specific low back pain (CNSLBP). Both healthy subjects and patients with CNSLBP will be randomized into three groups: one group will receive feedback from motion sensors, one group from a mirror and one group will receive no feedback (control group). A single session intervention with measurements at baseline and immediately post-intervention will be used.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific low back pain
* Age 18-65
* Able to understand Dutch

Exclusion Criteria:

* Subjects that received lumbar stabilization exercises in the past year
* Spinal surgery in the past
* Pregnancy
* Serious underlying pathologies (e.g. multiple sclerosis, tumors,…)
* Signs or symptoms of nerve root involvement
* Any physical condition at the moment of testing that can interfere with activities of daily living (e.g. serious knee pain)
* Known skin-allergy for tape
* BMI > 30kg/m²

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in lumbopelvic kinematics from baseline to immediately post-intervention | Day 1, immediately post-intervention
  Kinematics will be assessed using motion sensors that are mounted on the skin at the spinous processes of L1 and S1, and at the femur.

SECONDARY OUTCOMES:
usefulness of feedback (Numeric rating scale 0-10) | Day 1, immediately post-intervention
  How useful was the feedback that was provided to the subjects during the exercise trials?
Pain during the exercise trials (Numeric rating scale 0-10) | Day 1, immediately post-intervention
  Outcome measure primarily used as possible covariate
Fear of low back pain during the exercise trials (Numeric rating scale 0-10) | Day 1, immediately post-intervention
  Outcome measure primarily used as possible covariate
Fear of damaging the lumbar spine during the exercise trials (numeric rating scale 0-10) | Day 1, immediately post-intervention
  Outcome measure primarily used as possible covariate
Borg-scale to measure fatigue during the exercise trials | Day 1, immediately post-intervention
  Outcome measure primarily used as possible covariate

CONTACTS AND LOCATIONS:
Overall Officials: Annick Timmermans, prof. dr., Principal Investigator — Hasselt University; Enzo Olivieri, dr., Study Chair — Jessa Ziekenhuis, Hasselt, Belgium
Locations (2):
- Belgium (2):
  - Universiteit Hasselt, Diepenbeek
  - Jessa Ziekenhuis, Hasselt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Matheve T, Timmermans A, Danneels L, De Baets L. Task-Specific Perceived Harmfulness Predicts Protective Movement Behaviour in Chronic Low Back Pain. J Clin Med. 2024 Aug 25;13(17):5025. doi: 10.3390/jcm13175025. PMID 39274238
- [Derived] Matheve T, Brumagne S, Demoulin C, Timmermans A. Sensor-based postural feedback is more effective than conventional feedback to improve lumbopelvic movement control in patients with chronic low back pain: a randomised controlled trial. J Neuroeng Rehabil. 2018 Sep 26;15(1):85. doi: 10.1186/s12984-018-0423-6. PMID 30253807